CLINICAL TRIAL: NCT00792831
Title: Open Label, Uncontrolled, Pilot, Phase II Study of ITF2357 Administered Orally to Subjects With Chronic Lymphocytic Leukemia (CLL) Refractory/Relapsed After Conventional Chemotherapy or Relapsed After Autologous Bone Marrow Transplantation
Brief Title: Phase II Study of Histone-deacetylase Inhibitor ITF2357 in Refractory/Relapsed Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol needs complete restructuring in order to make it feasible and to complete the enrollment of 23 patients.
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/06/2357/21; 2006-005465-19 (EudraCT Number)
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — givinostat hydrochloride; givinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITF2357 (Experimental): ITF2357 was supplied as hard gelatine capsules for oral administration at the strength of 100 or 50 mg. Patients had to receive ITF2357 100 mg x 2/die at 12-hour intervals, in fed conditions, for three consecutive months.
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — Histone-Deacetylase Inhibitor
  Other Names: Givinostat

SUMMARY:
Primary objective:

- To determine overall response-rate, complete response (CR) or partial response (PR)

Secondary objectives:

* To assess the safety and tolerability of ITF2357;
* to assess total rate of responders (complete + partial responders);
* to determine the 6 months progression free survival;
* to determine the effects of the drug on haematological parameters.

DETAILED DESCRIPTION:
This is an open label, un-controlled, phase II, pilot clinical trial testing ITF2357 in a population of CLL patients relapsed after or refractory to conventional chemotherapy or relapsed after autologous bone marrow transplantation.

Patient received ITF 2357 orally at the dose of 100 mg x 2/die for three months with subsequent dose modifications if requested by the patient's conditions.

The study was prematurely discontinued due to recruitment problems. Since February 2008, date of first patient's first visit, until April 2009, date of early study discontinuation, only 3 patients were enrolled. The Sites involved in the study were 6 but only two actively recruited patients.

CLL is the most frequent type of leukemia in the western world and affects mainly elderly individuals, although about one third of patients are less than 60 years of age at diagnosis.

CLL is a heterogeneous disease characterised by a surprisingly diverse clinical course with patients that may have an overall survival time ranging from months to decades.

CLL accounts for approximately 7000 new cases and 4500 deaths per year in the US.

Chemotherapeutic treatment of CLL is largely ineffective and despite new emerging therapies, CLL still remains an incurable disease.

ITF 2357 is a novel and proprietary molecule synthesized by Italfarmaco S.p.A. Research Laboratories, provided with an established and powerful HDAC-inhibitory activity (see below for further details). It is being developed for a range of possible clinical applications both in oncohaematological conditions and in chronic inflammatory diseases. The former application is consistent with the well known antitumor pharmacological properties of HDAC-inhibitors as a family (i.e. cell-cycle arrest, pro-apoptotic and cell-differentiating effects); the latter application (chronic inflammation) is based of the demonstrated anticytokine effect of ITF 2357.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL according to the NCI Working Group criteria.
* Male and female patients of age >18 and ≤75 years
* Patients relapsed/refractory within 1 month after conventional chemotherapy (>1 polychemotherapy regimen) or relapsed within 3 months after autologous bone marrow transplantation
* ECOG performance score of ≤2
* Lymphocytes ≥10.0x10^9/L and platelets >75.0x10^9/L after recovery from a previous therapy
* Percentage of CD19+/CD5+ leukemic cells >50%
* Adequate cardiac, pulmonary and renal function, as defined by LVEF >45%, FEV >50% and creatinine ≤1.5 ULN or creatinine clearance ≥50ml/min
* Serum bilirubin <1.5xULN, AST and ALT <2.5xULN
* Serum potassium, phosphorus, total calcium, magnesium >LLN
* Normal values for FT4 and TSH (patients may be on thyroid hormone replacement)
* Negative test for beta-HCG for women in fertile age
* Documentation of written informed consent to participate in the trial
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Patients with Autoimmune haemolytic anaemia, Autoimmune Thrombocytopenic Purpura and Fischer Evans Syndrome.
* Patients with other autoimmune diseases.
* Patients with a marked baseline prolongation of QTc interval (e.g. repeated demonstration of a QTc interval >450 ms).
* Patients with history of additional risk factors for torsade de pointes (e.g. hearth failure, family history of Long QT Syndrome)
* The use of concomitant medications with potential risk of torsade de pointes and/or that can prolong QTc interval
* Prior treatment with an HDAC inhibitor.
* Treatment with Rituximab or Alemtuzumab within 90 days prior to study therapy.
* Patients HIV positive, patients with active EBV, HBV, HCV infection or liver cirrhosis
* Patients with active uncontrolled viral or bacterial or mycotic infection.
* Major surgeries within 4 weeks from study start or not fully recovered from any previous surgical procedure.
* Presence of any medical or psychiatric condition which may limit full compliance with the study or increase the risk associated with study participation or study drug administration.
* Patients in treatment with corticosteroids within 1 month before study start
* Significant cardiovascular disease (i.e., uncontrolled arrhythmias, unstable angina), or a major thromboembolic event (myocardial infarction, stroke, transient ischemic attack, pulmonary embolism, or non-catheter-related deep-vein thrombosis) in the last 6 months.
* Uncontrolled hypertension.
* Malabsorption syndromes.
* Breast feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Rate of complete response (CR) or partial response (PR) to ITF2357 in all patients | 13 weeks
  ITF2357 was given at 100 mg x 2/die for up to three months. A positive response was defined to be a patient experiencing a complete or partial remission.
  Complete remission (CR) Absence of lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms.
  Normal blood count: neutrophils ≥1.5x109/L, platelets >100x109/L, lymphocytes ≤4.0x109/L, Hb >11.0 g/dL (not supported by transfusion), BM biopsy: normal cellularity, lymphocytosis <30%.
  Partial remission (PR)
  ≥50% reduction in blood lymphocytes and ≥50% reduction in lymphadenophaty and/or 50% reduction in hepatomegaly and/or splenomegaly. Neutrophils ≥1.5x109/L or 50% improvement over baseline, platelets >100x109/L or 50% improvement over baseline, Hb >11.0 g/dL or 50% improvement over baseline (not supported by transfusion) It was considered PR
  * CR with nodular infiltrates at bone marrow biopsy (RPn)
  * CR with persistent anemia and thrombocytopenia therapy-related

SECONDARY OUTCOMES:
Total rate of responders (complete+partial responders) | 13 weeks
  ITF2357 was given at 100 mg x 2/die for up to three months
Six months progression free survival. | Up to 6 months
  ITF2357 was given at 100 mg x 2/die for up to three months
Number of subjects experiencing an adverse vents (AE), type, frequency, severity, timing and relatedness of AE | Throughout the study till 90 days post treatment
  ITF2357 was given at 100 mg x 2/die for up to three months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Martelli, MD, Study Director — Department of Internal Medicine and Public Health, University of Perugia
Locations (1):
- Department of Internal Medicine and Public Health, University of Perugia, Perugia, Italy